CLINICAL TRIAL: NCT03083717
Title: Application of Nanotechnology and Chemical Sensors for Diagnosis of Decompensated Heart Failure by Respiratory Samples
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Manhal Habib MD, PhD, Principal investigator, Rambam Health Care Campus
Other Study IDs: NaNose-CHF-2017
Record Dates: First submitted 2017-02-02; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with compensated heart failure
  Interventions: Diagnostic Test: Collection of breath samples, followed by analysis of exhaled breath using nanomaterial-based sensors (NaNose)
- Patients with decompensated heart failure
  Interventions: Diagnostic Test: Collection of breath samples, followed by analysis of exhaled breath using nanomaterial-based sensors (NaNose)
- Healthy subjects
  Interventions: Diagnostic Test: Collection of breath samples, followed by analysis of exhaled breath using nanomaterial-based sensors (NaNose)

INTERVENTIONS:
Diagnostic Test: Collection of breath samples, followed by analysis of exhaled breath using nanomaterial-based sensors (NaNose) — 2-3 liters of breath sample will be collected in chemically inert Mylar bags. The breath samples will then be immediately transferred from the Mylar bags to Tenax sorbent tubes using a dedicated pump. Tubes will be sealed and kept in 4˚C until NA-NOSE analysis.

SUMMARY:
Application of Nanotechnology and Chemical Sensors for Diagnosis of Decompensated Heart Failure by Respiratory Samples.

Breath testing, which links specific volatile molecular biomarkers in exhaled breath to medical conditions, is becoming increasingly popular as a non-invasive and potentially inexpensive diagnostic method for various diseases. NA-NOSE performs odor detection from exhaled breath, thus producing a distinct fingerprint for each mixture of analytes.

Several studies have been published, stating the advantages of these sensors, leading to promising outcomes in several fields.

The NA-NOSE breath test would be fast (examination and results would be obtained within 5-10 min), inexpensive, eventually portable (smaller than desktop computer), non-invasive and free of any side effects.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* ≥ 18 years of age, male or female
* Left ventricular Ejection fraction less than 40% or known to suffer from heart failure with preserved ejection fraction
* In decompensated heart failure group: dyspnea with confirmation of pulmonary congestion/edema by chest x-ray

Exclusion Criteria:

* Pericardial diseases, e.g. constrictive pericarditis, tamponade
* Significant congenital heart disease, up to the investigator's opinion
* Life-threatening or uncontrolled arrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or flutter with a resting ventricular rate >110 beats per minute.
* Acute ST elevation myocardial infarction
* Pregnant women
* Patients with pulmonary embolism
* Probable alternative diagnoses that in the opinion of the investigator could account for patient's HF symptoms (i.e., dyspnea), such as:

  1. significant pulmonary disease
  2. anemia with hemoglobin <10 g/dl
* participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from compensated heart failure (stable) Patients with decompensated acute heart failure Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-04-20 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of volatile organic compounds in breath samples | Each participant's breath sample will be analysed within one week of collection.
  Exhaled breath samples will be collected from each volunteer for characterization and identification using two different methods. The first method uses gas chromatography linked to mass spectrometry to identify and quantify the various breath volatile organic compunds (VOC's) in each group studied (compensated heart failure, decompensated heart failure and healthy subjects). The second method deploys cross-reactive nanoarrays in combination with pattern recognition methods (NaNose Technology).

CONTACTS AND LOCATIONS:
Overall Officials: Manhal A Habib, MD, PhD, Principal Investigator — Attending physician, Cardiology Unit, Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No